CLINICAL TRIAL: NCT04799106
Title: A Pilot Feasibility Study of Community Based Strategies for Early Detection of Melanoma
Brief Title: Community Based Strategies for Early Detection of Melanoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Robert Haile, Director, Cancer Research Center for Health Equity, Cedars-Sinai Medical Center
Other Study IDs: STUDY00001181
Record Dates: First submitted 2021-03-09; First posted 2021-03-16 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Community Based Strategies for Early Detection of Melanoma — The main procedures of this study include educational sessions about melanoma and how to detect it at its earliest stages with the help of a community health worker, conducting a self-skin examination every three months, helping to perform a skin examination every three months for a family member or friend who would be selected as a "partner", and completing short questionnaires at the beginning of the study, at month three during the study, and at completion of the study.

SUMMARY:
The purpose of this study is to pilot the use of community education and digital dermatology to increase the early detection of curable melanomas.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* >1mm lesion thickness with ulceration (T2b) or >2mm lesion thickness (T3/T4)
* Low socioeconomic status (SES) Non-Latinx White individuals (according to Yost's index SES level based on a principal components analysis)
* Latinx individuals
* Individual resides in semi-rural area, including zip codes within Antelope Valley in Southern California and Salinas in Northern California
* Individual speaks and reads English or Spanish
* Voluntary willingness and comprehension to consent

Exclusion Criteria:

Exclusion criteria is stage 0, I, IV, or unstaged diagnosis, or any individual who does not meet the above stated eligibility criteria will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 melanoma survivors drawn from the California Cancer Registry will be invited to participate in the study. Assuming a 20% response rate, approximately 40 individuals will be identified to participate in the study, including 20 in Southern California and 20 in Northern California. Participants will be invited to identify up to four friends or first-degree family members to also participate in the study, for a total of 200 participants.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Completion of self and partner skin examinations | 3 months
  Proportion of individuals recruited to those that follow through with the protocol
Completion of self and partner skin examinations | 6 months
  Proportion of individuals recruited to those that follow through with the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Robert Haile, DrPH, MPH, Principal Investigator — Cedars-Sinai